CLINICAL TRIAL: NCT01921894
Title: A Phase I Trial for Children With Vitamin D Insufficiency and High Risk of Severe Asthma Exacerbations
Brief Title: Vitamin D and Severe Asthma Exacerbations
Acronym: SAVED-P
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Juan Celedon, MD, MD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SAVED-P
Record Dates: First submitted 2013-08-09; First posted 2013-08-13 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-02

CONDITIONS: Asthma
Keywords: asthma; vitamin D
MeSH Terms: conditions — Asthma | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cholecalciferol 4000 IU (Experimental): Cholecalciferol 4000 IU oral chewable tablet once daily for 8 weeks
  Interventions: Dietary Supplement: Cholecalciferol
- Cholecalciferol 2000 IU (Experimental): Cholecalciferol 2000 IU oral chewable tablet once daily for 8 weeks
  Interventions: Dietary Supplement: Cholecalciferol
- Cholecalciferol 200 IU (Active Comparator): Cholecalciferol 200 IU oral chewable tablet once daily for 8 weeks
  Interventions: Dietary Supplement: Cholecalciferol

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — vitamin D supplementation with either 2,000 IU/day or 4,000 IU/day compared to vitamin D3 supplementation with 200 IU/day.
  Other Names: vitamin D3

SUMMARY:
This study of vitamin D is designed to assess both the safety and efficacy of potential doses (2,000 IU/day and 4,000 IU/day) in raising a vitamin D level to a normal range in a short period of time (e.g. 4 weeks or less) compared to 200 IU/day.

In children with vitamin D insufficiency or deficiency who are at risk for severe asthma exacerbations, we hypothesize that both vitamin D supplementation with 4,000 IU/day and 2,000 IU/day will safely achieve normal vitamin D levels, but that the higher dose (4,000 IU/day) will result in a larger proportion of subjects achieving this level at 4 and 8 weeks.

DETAILED DESCRIPTION:
Asthma is a major public health problem in the United States and worldwide. Severe disease exacerbations account for the majority of costs attributable to asthma in the United States. Vitamin D is an essential nutrient with significant immuno-modulatory effects. The observation that vitamin D insufficiency and asthma share risk factors such as urban residence, obesity, and African American ethnicity has generated significant interest in exploring a link between these two conditions.

This is an 8-week randomized, double-masked, controlled trial of vitamin D3 (2,000 IU/day and 4,000 IU/day) to achieve vitamin D sufficiency (a serum 25(OH)D ≥30 ng/ml in 60 school-aged children (ages 6 to 14 years) who have vitamin D insufficiency (a serum 25(OH)D <30 ng/ml) and are at risk for severe asthma exacerbations, but whose asthma that is well-controlled on medium-dose inhaled corticosteroid (ICS) at the end of a 4-week run-in period.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 6 years of age and younger than 15 years of age
* Have physician-diagnosed asthma
* Taking a medium dose of ICS (e.g. fluticasone 220mcg BID) for daily asthma control for at least 6 months in the prior year.
* Have had a severe asthma exacerbation in the previous year, defined as an Emergency Department (ED) visit, hospitalization, or unscheduled clinic visit for asthma resulting in intramuscular, intravenous, or oral steroids.
* Have bronchodilator responsiveness (BDR, an increase in FEV1 ≥12% from baseline after administration of inhaled albuterol) or (if no BDR) increased airway responsiveness to methacholine challenge
* Have vitamin D insufficiency (a serum vitamin D (25(OH)D) level <30 ng/ml)
* Have his/her parents give voluntary written consent to participate in the study

Exclusion Criteria:

* Chronic respiratory disorder other than asthma (e.g., bronchiectasis).
* Severe asthma, as evidenced by any of the following: a) chronic need for medication other than single controller therapy and inhaled β2-agonist, b) intubation for asthma at any time, and c) ≥2 hospitalizations or ≥6 severe asthma exacerbations in the previous year
* History of cigarette smoking in the prior year or former smoking if ≥5 pack-years
* Hepatic or renal disease, metabolic rickets, malabsorptive disorders, or other chronic diseases that would affect vitamin D metabolism
* Immune deficiency, cleft palate or Down's syndrome, which might increase the child's likelihood of respiratory infections
* Treatment with anticonvulsants or pharmacological doses of vitamin D (≥1,000 IU/day of vitamin D2 or D3)
* Chronic oral corticosteroid therapy
* Inability to perform acceptable spirometry
* Use of investigational therapies or participation in clinical trials 30 days before or during the duration of the study
* Serum calcium >10.8 mg/dl
* Serum 25(OH) D <10 ng/ml (severe vitamin D deficiency)

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2013-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Celedon, M.D., Dr.P.H., Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from: 1) the Emergency Department of Children's Hospital of Pittsburgh (CHP), 2) the Pulmonary Medicine and Allergy clinics of CHP, 3) the General Pediatric Clinics of CHP, and 4) participants in a prior study of the Pediatric Environmental Medicine Center of CHP (who had consented to be contacted about studies of asthma).
Pre-assignment Details: We recruited 48 children who met initial inclusion/exclusion criteria. Of these 48 children, 20 were excluded because of a 25(OH)D ≥30 ng/ml (n=13) or lack of bronchodilator response or airway responsiveness (n=7) at visit 1. Of the 28 remaining children, 4 were excluded because of non-adherence or poor asthma control during the run-in period.
Period: Overall Study
Arm/Group | Cholecalciferol 4000 IU | Cholecalciferol 2000 IU | Cholecalciferol 200 IU
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cholecalciferol 4000 IU | Cholecalciferol 2000 IU | Cholecalciferol 200 IU | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 8 | 8 | 24
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 2 | 11
  Male | 4 | 3 | 6 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic white | 2 | 2 | 5 | 9
  Non-Hispanic Black | 6 | 6 | 2 | 14
  Hispanic/Others | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sufficient Vitamin D Levels (≥30 ng/ml) After 8 Weeks of Supplementation
Description: The primary outcome of the proposed trial will be a sufficient (≥30 ng/ml) vitamin D level after 8 weeks of supplementation
Time Frame: 8 weeks
Population: In this pilot study, we wanted to report and compare the proportion of subjects who achieved vitamin D sufficiency after 8 weeks of treatment with one of three vitamin D doses.
Measure: Number; unit: participants
Groups:
- Cholecalciferol 4000 IU: All participants randomized to 4000 IU per day were analyzed. Outcome was defined as having vitamin D ≥30 ng/ml after 8 weeks.
- Cholecalciferol 2000 IU: All participants randomized to 2000 IU per day were analyzed. Outcome was defined as having vitamin D ≥30 ng/ml after 8 weeks.
- Cholecalciferol 200 IU: All participants randomized to 200 IU per day were analyzed. Outcome was defined as having vitamin D ≥30 ng/ml after 8 weeks.
Arm/Group | Cholecalciferol 4000 IU | Cholecalciferol 2000 IU | Cholecalciferol 200 IU
Number analyzed (Participants) | 8 | 8 | 8
participants | 8 | 6 | 4

2. Secondary Outcome: Number of Participants With Vitamin D Toxicity
Description: Participants with vitamin D toxicity, hypercalcemia (>10.8mg/dl) and/or an elevated urine Ca/Cr ratio (>0.37)
Time Frame: 8 weeks
Population: We wanted to report and compare the proportion of subjects who had vitamin D toxicity, hypercalcemia or an elevated UCa/UCr ratio across the three treatment arms
Measure: Number; unit: participants
Groups:
- Cholecalciferol 4000 IU: All participants randomized to 4000 IU per day were analyzed. Outcome was defined as having vitamin D toxicity, hypercalcemia (>10.8 mg/dl) or elevated uCa/uCr (>0.37).
- Cholecalciferol 2000 IU: All participants randomized to 2000 IU per day were analyzed. Outcome was defined as having vitamin D toxicity, hypercalcemia (>10.8 mg/dl) or elevated uCa/uCr (>0.37).
- Cholecalciferol 200 IU: All participants randomized to 200 IU per day were analyzed. Outcome was defined as having vitamin D toxicity, hypercalcemia (>10.8 mg/dl) or elevated uCa/uCr (>0.37).
Arm/Group | Cholecalciferol 4000 IU | Cholecalciferol 2000 IU | Cholecalciferol 200 IU
Number analyzed (Participants) | 8 | 8 | 8
participants | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Elevated Urinary Calcium/Creatinine Ratio
Description: Elevated urinary calcium/creatinine ratio defined as UCa/UCr > 0.37 after either 4 weeks or 8 weeks of supplementation
Time Frame: 4 and/or 8 weeks
Population: We wanted to compare the proportion of subjects who had an elevated UCa/UCr ratio across the three groups in this pilot Phase I Study
Measure: Number; unit: participants
Groups:
- Cholecalciferol 4000 IU: All participants randomized to 4000 IU per day were analyzed. Outcome was defined as having urinary calcium/creatinine ratio > 0.37
- Cholecalciferol 2000 IU; Cholecalciferol 200 IU: All participants randomized to 2000 IU per day were analyzed. Outcome was defined as having urinary calcium/creatinine ratio > 0.37
Arm/Group | Cholecalciferol 4000 IU | Cholecalciferol 2000 IU | Cholecalciferol 200 IU
Number analyzed (Participants) | 8 | 8 | 8
participants | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With FEV1 < 80% of Predicted
Description: Forced expiratory volume in 1 second (FEV1) as percent predicted (with reference values used according to the child's age, gender and ethnicity).
Time Frame: 8 weeks
Population: We wanted to compare the proportion of subjects whose FEV1 % predicted fell below 80% predicted across the three arms in this pilot Phase I study.
Measure: Number; unit: participants
Groups:
- Cholecalciferol 4000 IU: All participants randomized to 4000 IU per day were analyzed. Outcome was defined having FEV1 < 80% of predicted
- Cholecalciferol 2000 IU: All participants randomized to 2000 IU per day were analyzed. Outcome was defined having FEV1 < 80% of predicted
- Cholecalciferol 200 IU: All participants randomized to 200 IU per day were analyzed. Outcome was defined having FEV1 < 80% of predicted
Arm/Group | Cholecalciferol 4000 IU | Cholecalciferol 2000 IU | Cholecalciferol 200 IU
Number analyzed (Participants) | 8 | 8 | 8
participants | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Vitamin D Sufficiency (Vitamin D ≥30 ng/ml) After 4 Weeks of Supplementation
Description: The outcome is defined as the number of participants with a sufficient (≥30 ng/ml) vitamin D level after 8 weeks of supplementation
Time Frame: 4 weeks
Population: The characteristics of the study population are the same as described for the other primary outcome (vitamin D sufficiency at 8 weeks)
Measure: Number; unit: participants
Groups:
- Cholecalciferol 4000 IU: All participants randomized to 4000 IU per day were analyzed. Outcome was defined as having vitamin D ≥30 ng/ml after 4 weeks.
- Cholecalciferol 2000 IU; Cholecalciferol 200 IU: All participants randomized to 2000 IU per day were analyzed. Outcome was defined as having vitamin D ≥30 ng/ml after 4 weeks.
Arm/Group | Cholecalciferol 4000 IU | Cholecalciferol 2000 IU | Cholecalciferol 200 IU
Number analyzed (Participants) | 8 | 8 | 8
participants | 6 | 7 | 4

ADVERSE EVENTS:
Groups:
- Cholecalciferol 4000 IU: All participants randomized to 4000 IU per day were analyzed. Outcome includes any report of adverse events.
- Cholecalciferol 2000 IU: All participants randomized to 2000 IU per day were analyzed. Outcome includes any report of adverse events.
- Cholecalciferol 200 IU: All participants randomized to 200 IU per day were analyzed. Outcome includes any report of adverse events.
Arm/Group | Cholecalciferol 4000 IU | Cholecalciferol 2000 IU | Cholecalciferol 200 IU
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes